CLINICAL TRIAL: NCT03505788
Title: A Multi-center, Randomized, Double-blind, Phase IV Clinical Trial on the Diuretic Effects of Acetazolamide in Patients With Decompensated Heart Failure and Volume OveRload
Brief Title: Acetazolamide in Decompensated Heart Failure With Volume OveRload (ADVOR)
Acronym: Advor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Wilfried Mullens, Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZOLCAR17001
Record Dates: First submitted 2018-03-28; First posted 2018-04-23 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Acute Decompensated Heart Failure; Volume Overload
MeSH Terms: conditions — Edema | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-dose loop diuretics+placebo (Placebo Comparator): * At the moment of randomization (day 1), oral loop diuretics are stopped and the patient receives IV loop diuretics at a dose equal to the double of his oral daily maintenance dose + 500 mg IV bolus of placebo.
  * If the patient still have signs of volume overload the next mornings (day 2 and day 3), the patient will receive IV loop diuretics at a dose equal to the oral daily maintenance dose + 500 mg IV bolus of placebo. It the patient has no sign of volume overload at these time points, the study treatment will be stopped.
  Interventions: Drug: Placebo
- high-dose loop diuretics+acetazolamide (Experimental): * At the moment of randomization (day 1), oral loop diuretics are stopped and the patient receives IV loop diuretics at a dose equal to the double of his oral daily maintenance dose + 500 mg IV bolus of acetazolamide.
  * If the patient still have signs of volume overload the next mornings (day 2 and day 3), the patient will receive IV loop diuretics at a dose equal to the oral daily maintenance dose + 500 mg IV bolus of acetazolamide. It the patient has no sign of volume overload at these time points, the study treatment will be stopped.
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — In the experimental group, the patient will receive the standard of care loop diuretics and acetazolamide
  Arms: high-dose loop diuretics+acetazolamide
Drug: Placebo — In the placebo group, the patient will receive the standard of care loop diuretics and the placebo
  Arms: high-dose loop diuretics+placebo

SUMMARY:
This clinical research study is being conducted in multiple hospitals in Belgium and approximately 519 patients with acute decompensated heart failure are expected to participate. Large-scale research shows that 90% of the physicians treat volume overload with high doses of loop diuretics. However, there is not a lot of scientific data available regarding the optimal doses of these diuretic medications. In addition, it is observed that a lot of people, treated with these drugs, are being readmitted to the hospital due to a new episode of heart failure. The hypothesis of this study is that the volume overload could be better treated when patients receive a combination of different types of diuretics. Additionally, the total dose of the administrated diuretics might be lower this way.

DETAILED DESCRIPTION:
This is a randomized, double blind study with 2 treatment groups. This means that the patients will be randomized to one of the two treatment groups by chance. Patients randomized to the first group will receive standard treatment with high doses of intravenous loop diuretics and a placebo. Patients randomized to the other treatment group will receive a combination of the same doses of loop diuretics and an additional diuretic, acetazolamide (Diamox®). All diuretics will be administered intravenously. It is expected that the patients of the treatment group with the combination therapy will have a faster reduction of their fluid overload. In consequence the treatment duration and total dose of diuretics administered will be shorter. Acetazolamide (Diamox®) is a diuretic that acts at a different location in the kidney compared to the loop diuretics. This mutual reinforcement will probably reduce the total dose and duration of the diuretics.

The study will start during the hospitalization and will last around 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained before any study assessment is performed
* Male or female patients 18 years of age or older
* An elective or emergency hospital admission with clinical diagnosis of decompensated HF with at least one clinical sign of volume overload (e.g. oedema (score 2 or more), ascites confirmed by echography or pleural effusion confirmed by chest X-ray or echography)
* Maintenance therapy with oral loop diuretics at a dose of at least 1 mg bumetanide or an equivalent dose for at least 1 month before hospital admission (Conversion: 1 mg bumetanide = 40 mg furosemide = 20 mg torsemide)
* Plasma NT-proBNP levels >1000 ng/mL or BNP levels >250 ng/mL at the time of screening.
* Assessed LVEF by any imaging technique; i.e. echocardiography, catheterization, nuclear scan or magnetic resonance imaging within 12 months of inclusion

Exclusion Criteria:

* Concurrent diagnosis of an acute coronary syndrome defined as typical chest pain in addition to a troponin rise above the 99th percentile and/or electrocardiographic changes suggestive of cardiac ischemia
* History of congenital heart disease requiring surgical correction
* History of a cardiac transplantation and/or ventricular assist device
* Systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg at the moment of admission
* Expected use of intravenous inotropes, vasopressors or nitroprusside during the study. Use of nitrates is allowed only if the patient's systolic blood pressure is >140 mmHg
* Estimated glomerular filtration rate <20 mL/min/1.73m² at screening
* Use of renal replacement therapy or ultrafiltration at any time before study inclusion
* Treatment with acetazolamide during the index hospitalization and prior to randomization
* Exposure to nephrotoxic agents (i.e. contrast dye) anticipated within the next 3 days
* Use of any non-protocol defined diuretic agent with the exception of mineralocorticoid receptor antagonists. Thiazides, metolazone, indapamide and amiloride should be stopped upon study inclusion. If patient is taking a combination drug including a thiazide-type diuretic, the thiazide-type diuretic should be stopped
* Current use of sodium-glucose transporter-2 inhibitors
* Subjects who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wiflried Mullens, MD PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg AV, Genk, Limburg, Belgium

REFERENCES:
- [Derived] Van den Eynde J, Martens P, Dauw J, Nijst P, Meekers E, Ter Maaten JM, Damman K, Filippatos G, Lassus J, Mebazaa A, Ruschitzka F, Dupont M, Mullens W, Verbrugge FH. Serum Chloride and the Response to Acetazolamide in Patients With Acute Heart Failure and Volume Overload: A Post Hoc Analysis From the ADVOR Trial. Circ Heart Fail. 2024 Oct;17(10):e011749. doi: 10.1161/CIRCHEARTFAILURE.123.011749. Epub 2024 Aug 22. PMID 39171394
- [Derived] Meekers E, Dauw J, Martens P, Dhont S, Verbrugge FH, Nijst P, Ter Maaten JM, Damman K, Mebazaa A, Filippatos G, Ruschitzka F, Tang WHW, Dupont M, Mullens W. Renal function and decongestion with acetazolamide in acute decompensated heart failure: the ADVOR trial. Eur Heart J. 2023 Oct 1;44(37):3672-3682. doi: 10.1093/eurheartj/ehad557. PMID 37623428
- [Derived] Verbrugge FH, Martens P, Dauw J, Nijst P, Meekers E, Augusto SN Jr, Ter Maaten JM, Damman K, Filippatos G, Lassus J, Mebazaa A, Ruschitzka F, Dupont M, Mullens W. Natriuretic Response to Acetazolamide in Patients With Acute Heart Failure and Volume Overload. J Am Coll Cardiol. 2023 May 23;81(20):2013-2024. doi: 10.1016/j.jacc.2023.03.400. PMID 37197845
- [Derived] Martens P, Dauw J, Verbrugge FH, Nijst P, Meekers E, Augusto SN Jr, Ter Maaten JM, Damman K, Mebazaa A, Filippatos G, Ruschitzka F, Tang WHW, Dupont M, Mullens W. Decongestion With Acetazolamide in Acute Decompensated Heart Failure Across the Spectrum of Left Ventricular Ejection Fraction: A Prespecified Analysis From the ADVOR Trial. Circulation. 2023 Jan 17;147(3):201-211. doi: 10.1161/CIRCULATIONAHA.122.062486. Epub 2022 Nov 6. PMID 36335479
- [Derived] Mullens W, Dauw J, Martens P, Verbrugge FH, Nijst P, Meekers E, Tartaglia K, Chenot F, Moubayed S, Dierckx R, Blouard P, Troisfontaines P, Derthoo D, Smolders W, Bruckers L, Droogne W, Ter Maaten JM, Damman K, Lassus J, Mebazaa A, Filippatos G, Ruschitzka F, Dupont M; ADVOR Study Group. Acetazolamide in Acute Decompensated Heart Failure with Volume Overload. N Engl J Med. 2022 Sep 29;387(13):1185-1195. doi: 10.1056/NEJMoa2203094. Epub 2022 Aug 27. PMID 36027559

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Acetazolamide
Started | 260 | 259
Completed | 257 | 254
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Acetazolamide | Total
Number analyzed (Participants) | 260 | 259 | 519
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.5 (8.8) | 77.9 (9.0) | 78.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 89 | 194
  Male | 155 | 170 | 325
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 256 | 258 | 514
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Ischaemic aetiology [Count of Participants; unit: Participants] | 113 | 119 | 232
Weight [Mean (Standard Deviation); unit: kg] | 84.4 (19.7) | 85.3 (23) | 84.8 (21.4)
Heart rate [Mean (Standard Deviation); unit: bpm] | 77 (18) | 79 (19) | 78 (18)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 127 (22) | 126 (20) | 127 (21)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 73 (13) | 72 (13) | 72 (13)
Congestion score [Median (Inter-Quartile Range); unit: units on a scale] — Congestion scores range from 0 to 10 and are defined as the sum of scores for the degree of edema (0 to 4), pleural effusion (0 to 3), and ascites (0 to 3).
  Higher scores indicate a worse condition.
  units on a scale | 4 [3 to 6] | 4 [3 to 5] | 4 [3 to 6]
Composite of volume assessment score - Edema [Count of Participants; unit: Participants] — Number of patients with trace oedema (score 1 - pitting disappears immediately) clear pitting oedema (score 2), visual deformation above ankle (score 3) or visual deformation above knee (score 4)
  Participants | 241 | 237 | 478
Composite of volume assessment score - Pleural Effusion [Count of Participants; unit: Participants] — Number of patients with minor pleural effusion (score 2 - non amendable for punction) or major pleural effusion (score 3 - amendable for punction)
  Participants | 143 | 130 | 273
Composite of volume assessment score - Ascites [Count of Participants; unit: Participants] — Number of patients with minor ascites (score 2) or major ascites (score 3)
  Participants | 25 | 21 | 46
Maintenance dose - furosemide equivalent [Median (Inter-Quartile Range); unit: mg] | 60 [40 to 100] | 80 [40 to 120] | 60 [40 to 100]
LVEF [Mean (Standard Deviation); unit: %] | 43 (15) | 43 (15) | 43 (15)
Proportion LVEF ≤ 40% [Count of Participants; unit: Participants] | 111 | 113 | 224
NT-proBNP [Median (Inter-Quartile Range); unit: pg/mL] | 6483 [3262 to 11839] | 5600 [3034 to 10100] | 6173 [3068 to 10896]
NYHA [Count of Participants; unit: Participants] — Class I: No symptoms of heart failure. Class II: Symptoms of heart failure with moderate exertion, such as ambulating two blocks or two flights of stairs.
  Class III: Symptoms of heart failure with minimal exertion, such as ambulating one block or one flight of stairs, but no symptoms at rest.
  Class IV: Symptoms of heart failure at rest.
  Participants
    II | 35 | 31 | 66
    III | 148 | 148 | 296
    IV | 77 | 80 | 157
Serum hemoglobin [Mean (Standard Deviation); unit: g/dL] | 11.9 (2.0) | 11.9 (2.0) | 11.9 (2.0)
Sodium [Mean (Standard Deviation); unit: mmol/L] | 140 (4) | 139 (4) | 139 (4)
Serum creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 1.5 [1.2 to 1.9] | 1.5 [1.2 to 2.0] | 1.5 [1.2 to 1.9]
eGFR [Median (Inter-Quartile Range); unit: mL/min/1.73m^3] | 38 [29 to 51] | 40 [30 to 52] | 39 [29 to 52]
eGFR < 60mL/min/1.73m^3 [Count of Participants; unit: Participants] | 215 | 209 | 424
Comorbidities - History of atrial fibrillation [Count of Participants; unit: Participants] | 189 | 187 | 376
Comorbidities - Diabetes [Count of Participants; unit: Participants] | 133 | 112 | 245
Comorbidities - Hypertension [Count of Participants; unit: Participants] | 207 | 182 | 389
Use of ACEi/ARB/ARNi [Count of Participants; unit: Participants] — Use of Angiotensin-converting enzyme inhibitors (ACEi)/Angiotensin receptor blockers (ARB)/Angiotensin Receptor-Neprilysin Inhibitor (ARNi)
  Participants | 140 | 130 | 270
Beta-blocker [Count of Participants; unit: Participants] | 212 | 207 | 419
MRA [Count of Participants; unit: Participants] | 103 | 113 | 216
ICD [Count of Participants; unit: Participants] | 41 | 38 | 79
CRT [Count of Participants; unit: Participants] | 25 | 36 | 61

OUTCOME MEASURES:

1. Primary Outcome: Successful Decongestion
Description: defined as the absence of signs of volume overload, within 3 days after randomization and with no indication for escalation of decongestive therapy.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acetazolamide
Number analyzed (Participants) | 259 | 256
Participants | 79 | 108

2. Secondary Outcome: Mortality
Description: All-cause mortality during the first 3 months after start of the study
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acetazolamide
Number analyzed (Participants) | 259 | 256
Participants | 31 | 39

3. Secondary Outcome: Hospital Readmission
Description: If a patient is readmitted to the hospital within 3 months, this data will be collected
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acetazolamide
Number analyzed (Participants) | 259 | 256
Participants | 45 | 47

4. Secondary Outcome: Length of Index Hospital Admission
Description: The time frame between hospital admission and discharge will be calculated
Time Frame: 3 months
Measure: Geometric Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo | Acetazolamide
Number analyzed (Participants) | 259 | 256
days | 9.9 [9.1 to 10.8] | 8.8 [8.0 to 9.5]

5. Secondary Outcome: EuroQoL Five Dimensions Questionnaire (EQ-5D)
Description: A questionnaire about the patients' quality of life will be performed at baseline, the morning of day 4, at any readmission, 3 months. The questionnaire is divided into 5 levels of severity with a score varying from 1 to 5. 1 indicates no problems and 5 indicates severe problems. The EQ-5D-5L health status, defined by the EQ-5D-5L descriptive system, are converted into a single index value (utility data). Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead.
Time Frame: at baseline, day 4 (or discharge), at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Acetazolamide
Number analyzed (Participants) | 258 | 259
score on a scale
  Baseline | 0.571 (0.027) | 0.546 (0.027)
  Day 4 (or discharge) | 0.688 (0.028) | 0.656 (0.028)
  3 months FU | 0.592 (0.028) | 0.546 (0.028)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from collection of ICF up until 3 months follow-up (3 months after intervention).
Arm/Group | Placebo | Acetazolamide
All-Cause Mortality (participants affected / at risk) | 31/259 | 39/256
Serious Adverse Events (participants affected / at risk) | 124/259 | 123/256
Other Adverse Events (participants affected / at risk) | 184/259 | 192/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=259) | Acetazolamide (N=256)
Cardiac disorders (Cardiac disorders) | 80 | 80
Renal and urinary disorders (Renal and urinary disorders) | 15 | 20
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 | 3
Endocrine disorder (Endocrine disorders) | 0 | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 4 | 5
General disorders and administration site conditions (General disorders) | 4 | 4
Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 1
Infections and infestations (Infections and infestations) | 22 | 25
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 | 3
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 | 3
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7
Nervous system disorders (Nervous system disorders) | 2 | 0
Product issues (Product Issues) | 1 | 0
Psychiatric disorders (Psychiatric disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Surgical and medical procedures (Surgical and medical procedures) | 2 | 0
Vascular disorders (Vascular disorders) | 8 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=259) | Acetazolamide (N=256)
Cardiac arrhythmia (Cardiac disorders) | 30 | 29
Decreased and nonspecific blood pressure disorders and shock (Cardiac disorders) | 14 | 20
Heart failure (Cardiac disorders) | 83 | 69
Hyperkaelemia (General disorders) | 19 | 14
Hypokaelemia (General disorders) | 38 | 60

LIMITATIONS AND CAVEATS:
1. Nearly all patients were white
2. Patients had a history of chronic heart failure and had been receiving long-term outpatient treatment with at least 40 mg of furosemide equivalent.
3. Patients in the two trial groups received similar loop diuretics.
4. The congestion score focused on the presence of edema in the lower limb, pleural effusion, and ascites - reflective of mainly extracellular volume overload
5. The trial design excluded use of SGLT2 inhibitors

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT03505788/Prot_SAP_000.pdf